CLINICAL TRIAL: NCT06129552
Title: Basal Instincts: Towards Better Understanding of Basal Cell Function in Chronic Rhinosinusitis With Nasal Polyps
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: S67788
Record Dates: First submitted 2023-10-26; First posted 2023-11-13 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-10

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — The remaining human tissue from the upper respiratory tract consisting of surgical resected nasal turbinates, nasal polyps, and sinus tissue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls
  Interventions: Procedure: Conchotomy, aesthetic nose surgery or functional endoscopic sinus operation
- CRSwNP patients
  Interventions: Procedure: Conchotomy, aesthetic nose surgery or functional endoscopic sinus operation
- AR patients
  Interventions: Procedure: Conchotomy, aesthetic nose surgery or functional endoscopic sinus operation

INTERVENTIONS:
Procedure: Conchotomy, aesthetic nose surgery or functional endoscopic sinus operation — Conchotomy involves the reduction or removal of hypertrophic nasal turbinates, aesthetic nose surgery is a surgical procedure that aims to enhance the appearance of the nose, while functional endoscopic sinus surgery is a minimally invasive procedure focused on treating sinus conditions by removing obstructions and improving sinus drainage.

SUMMARY:
During this project, the investigators want to explore in vitro changes in basal cells and the crosstalk with residing immune cells as potential pathogenic mechanisms in CRSwNP vs healthy controls by using surgically resected patient samples.

DETAILED DESCRIPTION:
The investigators want to use patient and healthy control samples to study/compare the following aspects in vitro:

1. Investigate differences in epithelial and basal cell functions and differentiation characteristics.
2. Characterize the differences in epithelial cell populations and gene expression patterns. Also include an AR subset, to see if changes are specific for CRSwNP or more general for type 2 inflammatory disease of the upper airways.
3. Investigate basal cell activation via different environmental triggers through TLR stimulation.
4. Look at the genetic imprinting of basal cells before and after being exposed to specific triggers.
5. Investigate whether the secreted proteins from basal cells are chemotactic for other cell populations.
6. Investigate the interaction between basal and regulatory T cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Males and females

Exclusion Criteria:

* CRSwNP
* AR
* Smoker, or < 1-year ex-smoker
* Underlying systematic pathology (Morbus Wegener or Churg Strauss Syndrome for example)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CRSwNP patients:
  Inclusion Criteria:
  * Patients over the age of 18
  * Males and females
  * Patient with symptoms of chronic rhinosinusitis
  * Presence of nasal polyps
  Exclusion Criteria:
  * AR
  * Smoker, or < 1-year ex-smoker
  * Patient with cystic fibrosis
  * Only the presence of an antrochoanal polyp
  * Underlying systematic pathology (Morbus Wegener or Churg Strauss Syndrome for example)
  AR patients:
  Inclusion criteria:
  * Patients over the age of 18
  * Males and females
  * Patients with AR symptoms
  Exclusion criteria:
  * CRSwNP
  * Smoker, or < 1-year ex-smoker
  * Underlying systematic pathology (Morbus Wegener or Churg Strauss Syndrome for example)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Functional differences between epithelial/basal cells from CRSwNP samples in comparison to healthy controls assessed with functional assays. | 12-24 months
  Multiple techniques and functional assays will be used to fully investigate the functional differences between epithelial/basal cells isolated from healthy and CRSwNP samples. The differences in barrier composition will be assessed through TEER measurements (Ω × cm2) and FD4 permeability assays (ng/ml). Moreover, barrier composition is investigated by examining differences in membrane markers and junction expression through immunofluorescence and RT-qPCR. Finally, primary isolated cells will be used to assess protein levels through immunostainings, flow cytometry, and Western blots.
Characterization of differences in gene expression profiles and epithelial populations in/between CRSwNP and healthy controls assessed with different sequencing techniques. | 9-18 months
  To characterize differences in gene expression, or identify specific genes/cell populations that can contribute to CRSwNP, scRNA-sequencing will be performed, as well as bulk RNA sequencing. Depending on these results, specific triggers or receptors that can contribute to CRSwNP will be investigated by stimulation experiments. Besides, the effect on epigenetic imprinting before and after stimulation by performing ATAC-sequencing or DNA methylation profiling will be studied as well.
Changes and interactions in the basal and regulatory T-cell axis between healthy and CRSwNP-isolated cells will be studied through co-culture experiments. | 9-18 months
  The interaction between basal and regulatory T cells in relation to homeostasis and regeneration, and how this might change or contribute in/to CRSwNP will be investigated by co-culturing these cells. This will be assessed through the analysis of the supernatants using the Olink platform to investigate cytokines etc. Besides, there will be bulk RNA sequencing to look at changes in gene expression, as well as proliferation and growth assays to see the effect of T cells on basal cells and vice versa. To look at functional changes we can asses different functional assays and techniques (see outcome 1).

CONTACTS AND LOCATIONS:
Locations (1):
- Peter Hellings, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No